CLINICAL TRIAL: NCT02240342
Title: Ovarian Rejuvenation: Regeneration of Ovarian Follicles in Women With Poor Ovarian Reserve by Autologous Transplantation of Bone Marrow Derived Progenitors Cells in Peripheral Blood. Pilot Study.
Brief Title: Bone Marrow Transplantation to Promote Follicle Recruitment in Poor Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Dr. Antonio Pellicer Martínez, Professor, Hospital Universitario La Fe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEOFOL2014
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Ovarian Reserve
Keywords: Ovarian reserve; Poor response; Follicle recruitment; Bone marrow transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Poor ovarian reserve women (Experimental)
  Interventions: Drug: Bone marrow transplant into ovarian artery

INTERVENTIONS:
Drug: Bone marrow transplant into ovarian artery — Bone marrow progenitors mobilized to peripheral blood, obtained by plasmapheresis and infused into the ovarian artery

SUMMARY:
Women delay maternity and, as a consequence, available oocyte number and their quality decrease (9-18% of all IVF patients). Different treatment protocols have been developed nevertheless none of them optimal: the number of oocytes retrieved depends on the present ones. New generation of oocytes and follicles has been defended by some authors and bone marrow seems to be involved. What seems crucial is the niche that produces paracrine signals able to activate dormant cells and to attract undifferentiated cells from other tissues (homing). This phenomenon has been described by our group in other human reproductive tissues like endometrium. The purpose of the study is to improve ovarian reserve in unfertile women with poor ovarian reserve by means of bone marrow protective capacity.

Bone marrow progenitor cells will be delivered into the ovarian artery allowing them to colonize ovarian niche.

The study hypothesis is that bone marrow progenitor cells will improve ovarian reserve differentiating themselves into germ cells or, more likely, stimulating the niche to activate dormant follicles.

ELIGIBILITY:
Inclusion Criteria:

* < or= 40 years old
* FSH<15UI/L
* poor ovarian response after controlled ovarian stimulation with conventional doses (<3 oocytes) or two episodes of poor ovarian response after ovarian stimulation with maximal doses even if young or normal ovarian reserve study.
* Antral follicle count>2
* >1 antral follicle in the perfused ovary
* AMH between 0,5 and 3pmol/L
* regular menstrual bleeding each 21-35 days
* To be candidate to autologous hematopoietic progenitors transplantation

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Ovarian reserve | 6 months
  Measured by FSH-LH, oestradiol, AMH, antral follicle count

SECONDARY OUTCOMES:
Ovarian response to controlled ovarian stimulation | 6 months
  Number of MII oocytes obtained

OTHER OUTCOMES:
Take home baby | 2 years
  healthy new born after controlled ovarian stimulation, ICSI and ET.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La fe, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Herraiz S, Romeu M, Buigues A, Martinez S, Diaz-Garcia C, Gomez-Segui I, Martinez J, Pellicer N, Pellicer A. Autologous stem cell ovarian transplantation to increase reproductive potential in patients who are poor responders. Fertil Steril. 2018 Aug;110(3):496-505.e1. doi: 10.1016/j.fertnstert.2018.04.025. Epub 2018 Jun 28. PMID 29960701
- [Derived] Herraiz S, Buigues A, Diaz-Garcia C, Romeu M, Martinez S, Gomez-Segui I, Simon C, Hsueh AJ, Pellicer A. Fertility rescue and ovarian follicle growth promotion by bone marrow stem cell infusion. Fertil Steril. 2018 May;109(5):908-918.e2. doi: 10.1016/j.fertnstert.2018.01.004. Epub 2018 Mar 22. PMID 29576341